CLINICAL TRIAL: NCT06953011
Title: The Effect of Preferred Music on Anxiety and Comfort Levels in Thyroidectomy Surgery: A Randomized Controlled Trial (RCT)
Brief Title: The Effects of Different Types of Music on Patients Undergoing Thyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Çiçek SARUHAN, Lecturer, Dicle University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DicleU-ASBF-NURSE-ÇS-01
Record Dates: First submitted 2025-04-18; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Thyroid
Keywords: Anxiety; Thyroidectomy; Music; Patient comfort
MeSH Terms: conditions — Thyroid Diseases; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two groups with a conventional therapy control group
Who Masked: Investigator
Masking Description: Randomization was performed to ensure that patients who met the inclusion criteria among those admitted to the clinic for thyroidectomy surgery had an equal chance of being selected for the study. In order to perform randomized sampling, a table of random numbers was obtained over the internet in the computer environment by specifying the number of samples. A lottery method was then used to assign patients to either the intervention or control groups. To prevent mutual influence, patients were hospitalized in separate rooms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- music group (Experimental): Patients were met within 1 hour preoperatively. Vital signs, pain scores, and blood glucose levels were checked, and the state anxiety scale was administered. Music was played through headphones and speakers for at least 20 minutes, according to the patient's preference for both type and metod of listening. The state anxiety scale was then applied again. Patients' questions were answered and they were encouraged to share any concerns. Patient's questions were answered, and they were encouraged to share any concerns. They were prepared for surgery and transferred to the operating room. On the day after surgery, patients were visited again. Vital signs, pain scores, and blood glucose levels were checked and the perianesthesia comfort questionnaire (PCQ) was administered.
  Interventions: Other: music application
- control group (No Intervention): Patients were met within 1 hour preoperatively. Vital signs, pain score, and blood glucose were checked, and state anxiety scale was administered. Patients' questions were answered, and they were encouraged to share any concerns. They were then prepared for surgery and transferred to the operating room. On the day after surgery, patients were visited again. Vital signs, pain scores, and blood glucose levels were checked, and the perianesthesia comfort questionnaire (PCQ) was administered.

INTERVENTIONS:
Other: music application — Patients were met within 1 hour preoperatively. Vital signs, pain score, blood glucose were checked and state anxiety scale was applied. Music was played through headphones and speakers for at least 20 minutes according to the type of music preferred by the patients and the preferred way of listening to music, and the state anxiety scale was applied again. Patients' questions were answered and they were encouraged to share any concerns. Patients were prepared for surgery and transferred to the operating room. Considering the patient's recovery from anesthesia, patients were visited again the day after surgery, vital signs, pain score, blood glucose were checked and the perianesthesia comfort questionnaire (PCQ) was applied.
  Arms: music group

SUMMARY:
This study was conducted to investigate the effect preoperative music interventions on anxiety and postoperative comfort level in patients.

DETAILED DESCRIPTION:
Objective: This study was conducted to investigate the effect of preoperative music interventions on anxiety and postoperative comfort levels in patients.

Design: A randomized controlled quasi-experimental design was used. Methods: This study was conducted in the general surgery clinic of a university hospital in Diyarbakır, Turkey. A total of 100 patients (47 in the intervention and 53 in the control group) participated in the study by randomization. Personal Information Form, hemodynamic parameters, and State-Trait Anxiety Inventory were used for data collection. The State part of the State-Trait Anxiety Inventory was re-administered to the intervention group after the music intervention. In the postoperative period, hemodynamic parameters of all patients in both groups were monitoredş and the Perianesthesia Comfort Questionnaire was administered. SPSS 25.0 software was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18-65,
* Hospitalized for 24 hours after surgery,
* without cognitive impairment
* consenting to participate

Exclusion Criteria:

* Individuals under the age of 18 and over the age of 65
* Individuals with cognitive impairment
* Individuals who declined to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-23 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Scale | six months
  This scale is grounded in the two-factor theory of anxiety and comprises two sections with a total of 40 items. The items include both direct statements, which reflect negative emotional states, and reverse statements, which reflect positive emotional states. The total score ranges from 20 to 80, with higher scores indicating greater levels of anxiety. The first section (Items 1-20) assesses state anxiety, evaluating how the individual feels at a given moment. Respondents are asked to select one of the following options: Not at all, A little, A lot, or Completely. The second section (Items 21-40) measures trait anxiety, reflecting how the individual generally feels over time. For each item, respondents choose from: Almost never, Sometimes, Very often, or Almost always. The scale is intended to measure anxiety experienced over the past six months.

SECONDARY OUTCOMES:
Perianesthesia Comfort Questionnaire (PCQ) | six months
  This scale comprises 24 items designed to assess patients' general thoughts, self-perceptions, and emotional states before and after surgical procedures. The items are formatted using a 6-point Likert scale, with response options ranging from 1 (Strongly Disagree) to 6 (Strongly Agree). A total of 12 items are positively worded (Items 1, 5, 6, 11, 14, 16, 18, 19, 20, 21, 23, and 24), while the remaining 12 items are negatively worded (Items 2, 3, 4, 7, 8, 9, 10, 12, 13, 15, 17, and 22). Negatively worded items are reverse-coded during the scoring process.For positively worded items, higher scores indicate greater comfort, whereas lower scores reflect decreased comfort. The total scale score ranges from 24 to 144. Scoring involves summing the reverse-coded negative items and the original scores of positive items. A higher total score reflects a higher level of perceived comfort, while a lower score indicates reduced comfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Dicle University Hospital General Surgery Clinic, Diyarbakır, Sur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No